CLINICAL TRIAL: NCT06360458
Title: Methylprednisolone as Adjunct to Endovascular Thrombectomy for Patients With Acute Ischemic Strokes With Large Infarct: a Multicenter, Randomized, Double-blind, Placebo-controlled Trial (MIRACLE)
Brief Title: Methylprednisolone Adjunctive to Endovascular Thrombectomy for Stroke
Acronym: MIRACLE
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Wan-Jin Chen (Other)
Responsible Party: Sponsor-Investigator, Wan-Jin Chen, Vice President of Fujian Medical University and Vice President of The First Affiliated Hospital of Fujian Medical University, First Affiliated Hospital of Fujian Medical University
Organization: First Affiliated Hospital of Fujian Medical University (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: MRCTA,ECFAH of FMU[2024]368-1
Record Dates: First submitted 2024-04-07; First posted 2024-04-11 (Actual); Last update posted 2025-12-03 (Actual); Status verified 2025-11

CONDITIONS: Acute Ischemic Stroke; Large Infarct Core
MeSH Terms: conditions — Ischemic Stroke | interventions — Methylprednisolone Hemisuccinate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Methylprednisolone sodium succinate group (Experimental)
- Placebo group (Placebo Comparator): Methylprednisolone sodium succinate simulant
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Methylprednisolone sodium succinate — Intravenous injection of methylprednisolone sodium succinate (Chongqing Lummy Pharmaceutical Co., Ltd., 40mg/bottle) with a dose of 2mg/kg (maximum dose of 160mg), once daily, for three consecutive days. The initial study drug will be administered as soon as possible after randomization. It is recommended that the initial study drug administrated before arterial access closure, but it should not be delayed more than 2 hours after arterial access closure.
Drug: Placebo — Intravenous injection of placebo (Chongqing Lummy Pharmaceutical Co., Ltd., 40mg/bottle) with a dose of 2mg/kg (maximum dose of 160mg), once daily, for three consecutive days. The initial study drug will be administered as soon as possible after randomization. It is recommended that the initial study drug administrated before arterial access closure, but it should not be delayed more than 2 hours after arterial access closure.
  Arms: Placebo group

SUMMARY:
The efficacy and safety of methylprednisolone in acute ischemic stroke patients with large infarct cores (ASPECTS score < 6 or infarct volume ≥50 mL) due to anterior circulation large vessel occlusion have not been clearly established. This is a multi-center, randomized, double-blind, placebo-controlled trial to investigate early combination therapy with methylprednisolone for reperfusion in acute large core infarction.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years.
* The time from onset to randomization was within 12 hours.
* Anterior circulation ischemic stroke was preliminarily determined according to clinical symptoms or imaging examination.
* Occlusion of the intracranial internal carotid artery, the M1- or M2-segment of the middle cerebral artery by confirmed by CT angiography (CTA), MR angiography (MRA), or digital subtraction angiography (DSA).
* Baseline National Institutes of Health Stroke Scale (NIHSS) ≥ 6.
* Baseline Alberta Stroke Program Early CT Score (ASPECTS) < 6 (based on non-contrast CT or MRI) and/or core infarct volume ≥ 50 ml (based on CTP with rCBF < 30%).
* Planned treatment with endovascular thrombectomy (EVT).
* Informed consent obtained from patients or their legal representatives.

Exclusion Criteria:

* Intracranial hemorrhage confirmed by cranial CT or MRI.
* mRS score > 2 before onset.
* Pregnant or lactating women.
* Allergic to contrast agents or glucocorticoids.
* Participating in other clinical trials.
* The artery is tortuous so that the thrombectomy device cannot reach the target vessel.
* Bleeding history (gastrointestinal and urinary tract bleeding) in recent 1 month.
* Chronic hemodialysis and severe renal insufficiency (glomerular filtration rate < 30 ml/min or serum creatinine > 220 umol/L [2.5 mg/ dL]).
* Life expectancy due to any advanced disease < 6 months.
* Follow-up is not expected to be completed.
* Intracranial aneurysm and arteriovenous malformation.
* Brain tumors with imaging mass effect.
* Systemic infectious disease.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 928 (Actual)
Dates: Start 2024-08-01 (Actual); Primary Completion 2025-09-30 (Actual); Study Completion 2030-06-30 (Estimated)

PRIMARY OUTCOMES:
All-cause mortality at 90 (±14) days | From randomization to 90 (±14) days
  Primary Efficacy Outcome. Defined as the number of any cause deaths observed divided by the number of subjects observed over the 90-day study period.

SECONDARY OUTCOMES:
Time from randomization to the occurrence of death from any cause at 90 (±14) days | From randomization to 90 (±14) days
  Secondary Efficacy Outcome; To evaluate death rate of the two treatment groups
mRS ordinal shift at 90 (±14) days (scores 5 and 6 are merged) | From randomization to 90 (±14) days
  Secondary Efficacy Outcome
Proportion of patients with mRS score 0 to 4 at 90 (±14) days | From randomization to 90 (±14) days
  Secondary Efficacy Outcome
Proportion of patients with mRS score 0 to 3 at 90 (±14) days | From randomization to 90 (±14) days
  Secondary Efficacy Outcome
Proportion of patients with mRS score 0 to 2 at 90 (±14) days | From randomization to 90 (±14) days
  Secondary Efficacy Outcome
Proportion of patients with mRS score 0 to 1 at 90 (±14) days or return to pre-stroke mRS score (for patients with pre-stroke mRS > 1) | From randomization to 90 (±14) days
  Secondary Efficacy Outcome
Midline shift at 48 hours | From randomization to 48 hours
  Secondary Efficacy Outcome
Proportion of patients with midline shift >5 mm within 48 hours after EVT | From randomization to 48 hours
  Secondary Efficacy Outcome
Relative hemispheric volume at 48 hours | From randomization to 48 hours
  Secondary Efficacy Outcome.
Net water uptake at 48 hours | From randomization to 48 hours
  Secondary Efficacy Outcome
Proportion of patients with decompressive craniectomy after EVT | From randomization until the date of discharge, an average of 1 week
  Secondary Efficacy Outcome
NIHSS score at 5-7 days or at early discharge | From randomization to 5-7 days ( or at early discharge)
  Secondary Efficacy Outcome
EQ-5D-5L VAS at 90 (±14) days | From randomization to 90 (±14) days
  Secondary Efficacy Outcome
Proportion of patients with symptomatic intracranial haemorrhage (SICH) within 48 hours after EVT | From randomization to 48 hours
  Primary Safety Outcome. Based on the modified Heidelberg Bleeding Classification.
Proportion of patients with any intracranial haemorrhage (ICH) within 48 hours after EVT | From randomization to 48 hours
  Secondary Safety Outcome. Based on the modified Heidelberg Bleeding Classification.
Proportion of patients with pneumonia | From randomization until the date of discharge, an average of 1 week
  Secondary Safety Outcome
Proportion of patients with gastrointestinal haemorrhage within 7 days after EVT | From randomization to 7 days
  Secondary Safety Outcome
Incidence of any complications | From date of randomization until the date of discharge, an average of 1 week
  Secondary Safety Outcome
Incidence of any (serious) adverse events | From randomization to 90 (±14) days
  Secondary Safety Outcome

OTHER OUTCOMES:
mRS ordinal shift at 1 year (scores 5 and 6 are merged) | From randomization to 1 year
  Tertiary Efficacy Outcome
Proportion of patients with mRS score 0 to 2 at 1 year | From randomization to 1 year
  Tertiary Efficacy Outcome
Proportion of patients with mRS score 0 to 1 at 1 year or return to pre-stroke mRS score (for patients with pre-stroke mRS > 1) | From randomization to 1 year
  Tertiary Efficacy Outcome
mRS ordinal shift at 5 years (scores 5 and 6 are merged) | From randomization to 5 years
  Tertiary Efficacy Outcome
Proportion of patients with mRS score 0 to 2 at 5 years | From randomization to 5 years
  Tertiary Efficacy Outcome
Proportion of patients with mRS score 0 to 1 at 5 years or return to pre-stroke mRS score (for patients with pre-stroke mRS > 1) | From randomization to 5 years
  Tertiary Efficacy Outcome
EQ-5D-5L VAS at 1 year | From randomization to 1 year
  Tertiary Efficacy Outcome
EQ-5D-5L VAS at 5 years | From randomization to 5 years
  Tertiary Efficacy Outcome

CONTACTS AND LOCATIONS:
Locations (99):
- China (99):
  - The First Affiliated Hospital of USTC, Hefei, Anhui
  - Hefei First People's Hospital, Hefei, Anhui
  - Taihe County People's Hospital, Taihe Chengguanzhen, Anhui
  - Yijishan Hospital of Wannan Medical College, Wuhu, Anhui
  - Anxi County Hospital, Anxi, Fujian
  - Anxi Hospital of Traditional Chinese Medicine, Anxi, Fujian
  - Fuqing City Hospital of Fujian, Fuqing, Fujian
  - Fuzhou University Affiliated Provincial Hospital, Fuzhou, Fujian
  - Union Hospital Affiliated to Fujian Medical University, Fuzhou, Fujian
  - The Second Affiliated Hospital of Fujian University of Traditional Chinese Medicine, Fuzhou, Fujian
  - Department of Neurology, First Affiliated Hospital Fujian Medical University, Fuzhou, Fujian
  - 900th Hospital of PLA Joint Logistic Support Force, Fuzhou, Fujian
  - Longyan First Affiliated Hospital of Fujian Medical University, Longyan, Fujian
  - Nanping First Hospital, Nanping, Fujian
  - Mindong Hospital, Ningde, Fujian
  - Ningde Municipal Hospital, Ningde Normal University, Ningde, Fujian
  - Putian University Affiliated Hospital, Putian, Fujian
  - The First Hospital of Putian City, Putian, Fujian
  - Quanzhou First Hospital Affiliated to Fujian Medical University, Quanzhou, Fujian
  - The 910th Hospital of the Joint Logistics Support Force of the Chinese PLA, Quanzhou, Fujian
  - The Second Affiliated Hospital of Fujian Medical University, Quanzhou, Fujian
  - Sanming First Hospital, Sanming, Fujian
  - Shaowu Municiple Hospital, Shaowu, Fujian
  - The First Affiliated Hospital of Xiamen University, Xiamen, Fujian
  - Zhongshan Hosipital Xiamen University, Xiamen, Fujian
  - 909th Hospital of PLA Joint Logistic Support Force, Zhangzhou, Fujian
  - Zhangzhou Municipal Hospital of Fujian Province, Zhangzhou, Fujian
  - Gansu Province Central Hospital, Lanzhou, Gansu
  - Sun Yat-sen Memorial Hospital, Sun Yat-sen University, Guangzhou, Guangdong
  - Maoming Hospital of Traditional Chinese Medicine, Maoming, Guangdong
  - Maoming people's hospital, Maoming, Guangdong
  - Shantou Central Hospital, Shantou, Guangdong
  - Affiliated Hospital of Guangdong Medical University, Zhanjiang, Guangdong
  - Central people' s hospital of zhanjiang, Zhanjiang, Guangdong
  - Red Cross Hospital of Yulin City, Yulin, Guangxi
  - Guangzhou First People's Hospital, Guangzhou, Guangzhou
  - The First People's Hospital of Qingzhen, Qingzhen, Guizhou
  - The First Affiliated Hospital of Hainan Medical University, Haikou, Hainan
  - The Second Affiliated Hospital of Hainan Medical University, Haikou, Hainan
  - Biyan People's Hospital, Bishui, Henan
  - Xihua People's Hospital, Wacheng Neighborhood, Henan
  - Zhoukou Centeral Hospital, Zhoukou, Henan
  - ZhuMaDian Centeral Hospital, Zhumadian, Henan
  - Zhumadian First People's Hospital, Zhumadian, Henan
  - The Central Hospital of Enshi Tujia And Miao Automomous Prefecture, Enshi, Hubei
  - Ezhou Central Hospital, Ezhou, Hubei
  - Qichun People's Hospital, Huanggang, Hubei
  - Huanggang Central Hospital, Huanggang, Hubei
  - Huangshi Central Hospital, Huangshi, Hubei
  - Yangtze University Affiliated Hospital, Jingzhou, Hubei
  - Jingzhou Hospital Affiliated to Yangtze University, Jingzhou, Hubei
  - Lichuan City Ethnic Traditional Chinese Medical Hospital, Lichuan, Hubei
  - Shiyan Hospital of Integrated Traditional and Western Medicine, Shiyan, Hubei
  - Shiyan Renmin Hospital, Shiyan, Hubei
  - Taihe Hospital Affiliated to Hubei University of Medicine, Shiyan, Hubei
  - The First People's Hospital of Tianmen in Hubei Province, Tianmen, Hubei
  - Wuhan Hankou Hospital, Wuhan, Hubei
  - The Central Hospital of Wuhan, Tongji Medical College, Huazhong University of Science and Technology, Wuhan, Hubei
  - Wuhan NO.1 Hospital, Wuhan, Hubei
  - Tongji hospital, Tongji medical college, Huazhong university of science and technology, Wuhan, Hubei
  - The Third People's Hospital of Hubei Province, Wuhan, Hubei
  - Wuhan University Renmin Hospital, Wuhan, Hubei
  - Zhongnan Hospital of Wuhan University, Wuhan, Hubei
  - The First people's Hospital of Jiangxia District, Wuhan, Hubei
  - Xiangyang Hospital of Traditional Chinese Medicine, Xiangyang, Hubei
  - Xiangyang No.1 People's Hospital, Hubei University of Medicine., Xiangyang, Hubei
  - Xianning Central Hospital, Xianning, Hubei
  - The Second People's Hospital of Yichang, Yichang, Hubei
  - Baotou Central Hospital, Baotou, Inner Mongolia
  - The Affiliated Hospital of Xuzhou Medical University, Xuzhou, Jiangsu
  - First Affiliated Hospital of Gannan Medical University, Ganzhou, Jiangxi
  - Ganzhou People's Hospital, Ganzhou (G.Z.), Ganzhou, Jiangxi
  - Jingdezhen First People's Hospital, Jingdezhen, Jiangxi
  - Jiujiang University Affiliated Hospital, Jiujiang, Jiangxi
  - The First People's Hospital of Jiujiang, Jiujiang, Jiangxi
  - Jiangxi Provincial People's Hospital, Nanchang, Jiangxi
  - The First Affiliated Hospital, Jiangxi Medical College, Nanchang University, Nanchang, Jiangxi
  - Yingtan people's hospital, Yingtan, Jiangxi
  - The First People's Hospital of Xianyang, Xianyang, Shaanxi
  - Affiliated Hospital of Shandong University of Traditional Chinese Medicine, Jinan, Shandong
  - Jinan Central Hospital Affiliated to Shandong First Medical University, Jinan, Shandong
  - Liaocheng People's Hospital, Liaocheng, Shandong
  - Liaocheng third people's hospital, Liaocheng, Shandong
  - The Affiliated Hospital of Qingdao Univercity, Qingdao, Shandong
  - The Second Affiliated Hospital of Shandong First Medical University, Tai’an, Shandong
  - Zoucheng People's Hospital, Shandong Province, Zoucheng, Shandong
  - Ruijin Hospital, Shanghai Jiaotong University School of Medicine, Shanghai, Shanghai Municipality
  - Cardiovascular Hospital Affiliated to Shanxi Medical University, Taiyuan, Shanxi
  - Shanxi Provincial People's Hospital, Taiyuan, Shanxi
  - Chongzhou People's Hospital, Chengdu, Sichuan
  - Gulin County People's Hospital, Gulin, Sichuan
  - Mianyang 404 Hospital, Mianyang, Sichuan
  - Mianyang Central Hospital, School of Medicine, University of Electronic Science and Technology of China, Mianyang, Sichuan
  - Affiliated Hospital of North Sichuan Medical College, Nanchong, Sichuan
  - Suining Central Hospital, Suining, Sichuan
  - Zigong Third People's Hospital, Zigong, Sichuan
  - Tianjin Huanhu Hospital, Tianjin, Tian
  - Bozhou People's Hospital, Bole, Xinjiang
  - Qujing NO.1 Hospital, Qujing, Yunnan

IPD SHARING:
Plan to Share IPD: No